CLINICAL TRIAL: NCT06214078
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, Parallel-group Clinical Trial of Nicotinamide Mononucleotide in the Treatment of Mild Ulcerative Colitis
Brief Title: Preliminary Clinical Study of NMN Intervention in Mild Ulcerative Colitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-NMN-XY3
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Ulcerative Colitis Chronic Mild
MeSH Terms: interventions — Nicotinamide Mononucleotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NMN group (Experimental): Patients in this group will take nicotinamide mononucleotide capsules orally twice daily for 8 weeks, one capsule per time, each actually containing 250mg of nicotinamide mononucleotide.
  Interventions: Dietary Supplement: nicotinamide mononucleotide
- placebo group (Placebo Comparator): Patients in this group will receive 1 placebo capsule orally twice daily for 8 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: nicotinamide mononucleotide — Nicotinamide mononucleotide (NMN), a bioactive substance found in a variety of foods, is a precursor for the synthesis of nicotinamide adenine dinucleotide (NAD+). NAD+ plays a crucial role in a variety of biological processes including cell death, senescence, gene expression, neuroinflammation, and DNA repair.
  Arms: NMN group
Other: placebo — The placebo mimicked the appearance and properties of nicotinamide mononucleotide(NMN) enteric-coated capsules. The specifications, usage and dosage of placebo were the same as those of NMN.
  Arms: placebo group

SUMMARY:
The goal of this clinical trial is to compare the safety and efficacy of nicotinamide mononucleotide (NMN) and placebo in patients with mild ulcerative colitis (UC). The main question it aims to answer is Whether NMN can alleviate the intestinal pathology of UC patients, so as to play a role in UC treatment or adjuvant therapy.

Participants will be randomized into two groups, an NMN group or a placebo group. Patients in the NMN group were treated with NMN intervention for 8 weeks. The placebo group received a placebo intervention for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, ≤75 years old;
2. Clinical diagnosis of mild active UC patients, the diagnosis standard reference inflammatory bowel disease diagnosis and treatment of the consensus of opinion 2018.
3. Agreed to participate in this study, and sign the informed consent.

Exclusion Criteria:

1. Patients with ALT or AST more than 2 times the upper limit of normal, TBIL more than 2 times the upper limit of normal;
2. The creatinine clearance patients less than 60 ml/min.
3. The intestines or other parts have severely active infection patients need to use antibiotics or antiviral drugs;
4. Crohn's disease and intestinal tuberculosis and other chronic intestinal infectious disease, intestinal malignant tumor patients;
5. Pregnancy and lactation women;
6. People with diabetes or screening period more than 7.0 tendency for fasting glucose/L or glycosylated hemoglobin exceed 6.5%;
7. With serious mental illness, such as drugs and alcohol can't cooperate with the patients;
8. Participated in any other clinical investigator within 1 month before the screening period;
9. The researchers determine any other disease or condition is not suitable for patients participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate | 8 weeks
  Clinical response was defined according to STRIDE II as a reduction of at least 50% in Patient Reported Outcomes 2 (PRO2) rectal bleeding and stool frequency.

SECONDARY OUTCOMES:
Biomarker target attainment rate | 8 weeks
  The target of inflammatory biomarkers was defined as normal C-Reactive Protein (CRP) + Fecal Calprotectin (FC) decreased to 100-250 ug/g.
clinical remission rate | 8 weeks
  It was defined as modified Mayo score ≤2 and no single subscore > 1.
Endoscopic remission rate | 8 weeks
  Endoscopic remission was defined as Mayo endoscopic score (MES) =0 or UCEIS score ≤1.
Histologic remission rate after 8 weeks of intervention | 8 weeks
  Histological remission: Geboes index score < 2.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Wang, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
Some data underlying this trial cannot be shared publicly due to protection of participant's privacy.